CLINICAL TRIAL: NCT05192967
Title: Development and Efficiency Evaluation of a Respiratory Disease Pandemics Preparedness Training Program for Pre-Hospital Emergency Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seval Çalışkan Pala (Other)
Responsible Party: Sponsor-Investigator, Seval Çalışkan Pala, Research Assistant Doctor, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EskisehirOU99
Record Dates: First submitted 2021-12-14; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: During the Pandemic Process the Focus is on Developing a Training Program

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1 (Experimental): The training program determined to the experimental group was applied with video. Training program content:
  1. Knowledge, attitude, skills about COVID-19
  2. Approach to the COVID-19 positive case
  3. Communication skills
  4. Psychological resilience
  Interventions: Behavioral: Pandemic preparedness via video
- Experimental 2 (Experimental): The training program determined to the experimental group was applied with video.
  Training program content:
  1. Knowledge, attitude, skills about COVID-19
  2. Approach to the COVID-19 positive case
  3. Communication skills
  4. Psychological resilience
  Interventions: Behavioral: Pandemic preparedness via video
- Control 1 (Other): The training program determined to the control group was applied with classical method.
  Training program content:
  1. Knowledge, attitude, skills about COVID-19
  2. Approach to the COVID-19 positive case
  3. Communication skills
  4. Psychological resilience
  Interventions: Behavioral: Pandemic preparedness via classical method
- Control 2 (Other): The training program determined to the control group was applied with classical method.
  Training program content:
  1. Knowledge, attitude, skills about COVID-19
  2. Approach to the COVID-19 positive case
  3. Communication skills
  4. Psychological resilience
  Interventions: Behavioral: Pandemic preparedness via classical method

INTERVENTIONS:
Behavioral: Pandemic preparedness via video — A training program created by experts on knowledge, attitude, skills, simulated case approach, communication between the patient and the team, and psychological resilience about COVID-19 was implemented with a video demonstration.
  Arms: Experimental 1; Experimental 2
Behavioral: Pandemic preparedness via classical method — A training program created by experts on knowledge, attitude, skills, simulated case approach, communication between the patient and the team, and psychological resilience about COVID-19 was implemented with a classical method.
  Arms: Control 1; Control 2

SUMMARY:
Pre-hospital emergency health workers, who are on the front line among healthcare workers, are at greater risk in epidemic situations, as they are the first team to come into contact with the patient and are responsible for making necessary interventions by staying in close contact with the patient during the transfer process (1, 2). Health workers need to improve their knowledge, attitudes and skills during the pandemic process; on the other hand, they experience mental and communicative problems more strikingly. It is essential to increase the continuity of development, mental resilience, and communication of healthcare professionals(3). A randomised controlled study was planned to prepare a training program to improve pre-hospital emergency health workers' knowledge, attitudes, and skills about pandemic preparations and evaluate its effectiveness.

The intervention study was conducted among pre-hospital emergency health workers in Eskişehir between July 2020 and December 2021. Ethics committee approval and administrative permissions were obtained. In the study, when the type 1 (α) error was 5%, and the type 2 error (1-β) was 95%, the effect size was accepted as 0.5, and it was calculated with the G*Power 3.1 statistical program that there should be at least 47 people in the groups. The study population consists of paramedics and emergency medical technicians(EMT) (N=420) in Eskişehir city, Turkey. Each participant in the study population was given a score by propensity score matching analysis according to age, gender, occupational group (paramedic and EMT), working time (year) variables. The study list was arranged according to the initials of their surnames, and the drawing method was used while assigning those with similar scores to four groups (experimental 1, experimental 2, control 1, control 2). Four groups, two interventions and two controls, were included in the study.

The work consisted of five stages:

1. Determining the needs in education,
2. Development of educational materials,
3. Making pre-training measurements,
4. Implementation of the training program,
5. Performing post-training measurements. As a result of the evaluation, the subjects that healthcare professionals need to train were determined as knowledge, attitude, skills, infection control measures, communication skills, psychological resilience and attitudes of healthcare professionals to the patient in a simulated case and pandemic. The appropriate data collection form was chosen after the training program's content was determined. Before the intervention, the first measurements were taken via the COVID-19 knowledge, attitude, skills, and perceived barriers to infection control questionnaire, the communication competence scale, the psychological resilience scale, and the data collection form, including the simulated case approach. After the training program's content was determined, training was given to the intervention group with a video screening and the control group with the classical training method. After the training program, a post-test was applied after a four-week follow-up.

DETAILED DESCRIPTION:
The intervention study was conducted among pre-hospital emergency health workers in Eskişehir between July 2020 and December 2021. Ethics committee approval and administrative permissions were obtained. In the study, when the type 1 (α) error was 5%, and the type 2 error (1-β) was 95%, the effect size was accepted as 0.5, and it was calculated with the G*Power 3.1 statistical program that there should be at least 47 people in the groups. The study population consists of paramedics and emergency medical technicians (N=420) in Eskişehir city, Turkey. Each participant in the study population was given a score by propensity score matching analysis according to age, gender, occupational group (paramedic and ATT), working time (year) variables. The study list was arranged according to the initials of their surnames, and the drawing method was used while assigning those with similar scores to four groups (experimental 1, experimental 2, control 1, control 2). Four groups, two interventions and two controls, were included in the study. The work consisted of five stages:

1. Determining the needs in education,
2. Development of educational materials,
3. making pre-training measurements,
4. Implementation of the training program,
5. Performing post-training measurements. As a result of the evaluation, the training needs of healthcare professionals were determined as knowledge, attitude, skills, infection control measures, communication skills, psychological resilience and approach to COVID-19 positive case. After the training program's content was determined, training was given to the intervention group with a video screening and the control group with the classical training method.

Measurement tools used in the study:

1. Questionnaire on knowledge, skills, attitudes and perceived barriers in infection control about COVID-19: Adapting the questionnaire named "Knowledge, attitude, practice and perception barriers among healthcare professionals regarding COVID-19", developed by Saqlain et al., into Turkish, and conducting a reliability and validity study It was made by Caliskan Pala et al. in 2021 (4, 5).
2. Simulated case checklist: It was created to evaluate the case approach of healthcare professionals during the pandemic process. The template of events for applied and critical healthcare simulation (Teach Sim) and The Simulation team assessment tool (STAT) created simulated cases. According to START, which is the most widely used triage system, a total of 111 cases were developed, with cases according to green, yellow, and red triage codes. (6). The approach of each participant to a COVID-19 positive case with a green code ( Minor injuries), one yellow ( Non-life-threatening injury ), and one red ( Life-threatening injury ) was evaluated. Each scenario consisted of six steps, 20 questions regarding infection control measures, patient history and physical examination, preliminary diagnosis, medical intervention, communication, and delivering the patient to the health institution. Each item on the scale was scored according to its completion status. The score that can be obtained according to the number of questions in the steps was standardised.
3. communication skills: This scale, which aims to measure the communication skills of individuals in general, was developed by Wiemann in 1977 and adapted into Turkish by Koca and Erigüç in 2017 (7, 8). The scale consists of eight sub-dimensions: "Social Behavior Competence", "Individual aspects in communication", "Empathy competency", "Adaptability", "Sensitivity Competence", "Communication Encouragement Competence", "Human Relations", "Listening Competence".
4. psychological resilience: The scale was developed by Friborg et al. in 2003, and Basım and Çetin established Turkish validity and reliability in 2011 (9, 10). The structural style consists of six sub-areas: future perception, family harmony, self-perception, and social competence.

Hypotheses:

1. Is the pandemic preparedness training program effective in developing knowledge, attitudes and skills in pre-hospital emergency health workers compared to the control group trained with the classical method?
2. Is the pandemic preparedness training program effective in developing communication competence in prehospital emergency health workers compared to the control group trained with the classical method?
3. Is the pandemic preparedness training program effective in developing psychological resilience in prehospital emergency health workers compared to the control group trained with the classical method?

ELIGIBILITY:
Inclusion Criteria:Being a pre-hospital emergency health worker(paramedic or EMT) -

Exclusion Criteria:not completing the stages of the study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitude, practice and perceived barriers among healthcare workers regarding COVID-19 Questionnaire | One month
Simulated case checklist | One month
Communication skills | One month
  Measurement was made with the communication competence scale
Psychological resilience | One month
  Measurement was made with the psychological resilience scale

CONTACTS AND LOCATIONS:
Overall Officials: Seval CALISKAN PALA, Study Director — ESOGU; Selma METİNTAS, Principal Investigator — ESOGU; Engin OZAKIN, Study Chair — ESOGU
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided